CLINICAL TRIAL: NCT02585635
Title: Risk Models to Optimise Prophylaxis Schedules in Children With Haemophilia
Acronym: MOrPH
Status: Completed | Type: Observational
Sponsor: Neuroscience Research Australia (Other)
Collaborators: Sydney Children's Hospitals Network (Other); The George Institute (Other); Royal Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: H15-263263
Record Dates: First submitted 2015-10-14; First posted 2015-10-23 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Families: Families of children with haemophilia
- Clinicians: Haemophilia physicians

SUMMARY:
The MOrPH study is designed to identify optimal prophylaxis schedules for children with haemophilia. This involves development of combined pharmacokinetic and pharmacodynamic models. Interpretation of model outputs will be informed by two surveys. The first will survey families of children with haemophilia to ascertain families' values and preferences concerning prophylaxis schedules. The second will survey haemophilia physicians to ascertain the criteria physicians use to prescribe prophylaxis schedules.

DETAILED DESCRIPTION:
Methods: Part I (surveys)

Two cross-sectional surveys will be conducted, a family survey and a clinician survey. The surveys will be completed online. Participation will be voluntary and anonymous.

Family survey. The family survey will identify preferences of families of children with haemophilia for different prophylaxis schedules. At least 20 families will participate. This number should provide a clear indication of family's preferences for different prophylaxis schedules.

People will be eligible to participate in the family survey if they have haemophilia A or B and are aged between 14 and 17 years, or if they are the parent of a child (< 18 years) with haemophilia.

Participants will be recruited using advertisements placed in community print-based and/or electronic communications and, if necessary, by inviting families attending a youth camp for people with haemophilia. The survey will ask participants about the characteristics of the child with haemophilia including the child's age, current level and frequency of physical activity and sports participation, current prophylactic medication schedule and method of administration. They will also be asked to rate the acceptability of a number of possible prophylactic schedules as "acceptable", "marginally acceptable" or "unacceptable".

Clinician survey. The second survey will be of physicians. To be eligible, participants must be physicians currently practising in paediatric haemophilia treatment centres. Participants will be asked to rank factors that influence their decision making when advising patients regarding prophylactic scheduling. These factors include: cost, tolerability for families, venous access, physical activity and sport, pharmacokinetics, inhibitor development and age. They will also be asked to report on which prophylactic schedules they would considerable unacceptable, putting aside issues regarding efficacy.

Methods: Part II (modelling)

The MOrPH project will use pharmacokinetic and pharmacodynamic modelling to identify optimal prophylaxis schedules. Conventional pharmacokinetic models will be used to identify prophylaxis schedules that maximise time above threshold and minimise trough values of clotting factor concentrates. In addition, pharmacodynamic models will be developed to provide child-specific predictions of the risk of bleeds as a function of prophylaxis schedules. The pharmacodynamic models will be used to identify prophylaxis schedules that minimise risk of bleeds.

ELIGIBILITY:
Inclusion Criteria:

* People will be eligible to participate in the family survey if they have haemophilia A or B and are aged between 14 and 17 years, or if they are the parent of a child (< 18 years) with haemophilia
* People will be eligible to participate in the physician survey if they are physicians currently practising in paediatric haemophilia treatment centres.

Exclusion Criteria:

* Unable to communicate effectively in English.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: There will be two study populations:
  1. Families of children with haemophilia
  2. Haemophilia physicians
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2016-03; Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Acceptability of injection frequencies | Day 1 (i.e. on the day of response to the survey)
  Families will be asked to rate as "acceptable", marginally acceptable" or "unacceptable" different frequencies of prophylactic factor injections.
Acceptability of time of injections | Day 1 (i.e. on the day of response to the survey)
  Families will be asked to rate as "acceptable", marginally acceptable" or "unacceptable" different injection times.
Importance of factors influencing prescription of prophylaxis schedules | Day 1 (i.e. on the day of response to the survey)
  Physicians will be asked to rank the importance of factors (including cost, tolerability for families, venous access, physical activity and sport, pharmacokinetics, inhibitor development and age) that influence their prescription of prophylaxis schedules.

CONTACTS AND LOCATIONS:
Overall Officials: Rob Herbert, PhD, Principal Investigator — Neuroscience Research Australia

IPD SHARING:
Plan to Share IPD: No